CLINICAL TRIAL: NCT00085644
Title: A Phase 3 Multicenter Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Active Ankylosing Spondylitis
Brief Title: Human Anti-tumor Necrosis Factor (TNF) Monoclonal Antibody Adalimumab in Subjects With Active Ankylosing Spondylitis
Acronym: ATLAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Laura Redden, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-607
Record Dates: First submitted 2004-06-10; First posted 2004-06-16 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental)
  Interventions: Biological: adalimumab (D2E7)
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab (D2E7) — Adalimumab 40 mg every other week, subcutaneous
  Other Names: ABT-D2E7; adalimumab; Humira
  Arms: Adalimumab
Biological: placebo — Placebo every other week, subcutaneous
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of adalimumab 40 mg given every other week (eow) in subjects with active ankylosing spondylitis (AS) who have had an inadequate response to, or who are intolerant to, treatment with at least 1 nonsteroidal anti-inflammatory drug (NSAID) and who may have also failed treatment with at least 1 disease-modifying antirheumatic drug (DMARD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >= 18 years of age
* meet Modified NY Criteria definition of ankylosing spondylitis (AS)
* have diagnosis of active AS based on protocol specified criteria
* inadequate response or intolerance to >= 1 nonsteroidal antiinflammatory drug (NSAID)
* be able and willing to learn to self-administer subcutaneous (SC) injections

Exclusion Criteria:

* Active tuberculosis, listeriosis,or hepatitis B, or any history of hepatitis C
* History of demyelinating disease, multiple sclerosis, cancer, or lymphoproliferative disease
* Previous anti-tumor necrosis factor therapy
* Treatment with disease-modifying antirheumatic drugs (DMARDs - other than methotrexate, hydroxychloroquine, and sulfasalazine)
* Treatment with intra-articular corticosteroid joint injections within 4 weeks of study dosing
* Biologic or investigational therapy within 6 weeks of study dosing
* Treatment with intravenous (IV) antibiotics within 30 days of study dosing
* Treatment with oral antibiotics within 14 days of study dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2004-01; Primary Completion 2004-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, PhD, Study Director — Abbott
Locations (21):
- United States (21):
  - Birmingham, Alabama
  - Mobile, Alabama
  - San Francisco, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Portland, Maine
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Albany, New York
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington

REFERENCES:
- [Derived] van der Heijde D, Breban M, Halter D, DiVittorio G, Bratt J, Cantini F, Kary S, Pangan AL, Kupper H, Rathmann SS, Sieper J, Mease PJ. Maintenance of improvement in spinal mobility, physical function and quality of life in patients with ankylosing spondylitis after 5 years in a clinical trial of adalimumab. Rheumatology (Oxford). 2015 Jul;54(7):1210-9. doi: 10.1093/rheumatology/keu438. Epub 2014 Dec 25. PMID 25541333
- [Derived] Kimel M, Revicki D, Rao S, Fryback D, Feeny D, Harnam N, Thompson C, Cifaldi M. Norms-based assessment of patient-reported outcomes associated with adalimumab monotherapy in patients with ankylosing spondylitis. Clin Exp Rheumatol. 2011 Jul-Aug;29(4):624-32. Epub 2011 Aug 31. PMID 21813060
- [Derived] Revicki DA, Rentz AM, Luo MP, Wong RL. Psychometric characteristics of the short form 36 health survey and functional assessment of chronic illness Therapy-Fatigue subscale for patients with ankylosing spondylitis. Health Qual Life Outcomes. 2011 May 22;9:36. doi: 10.1186/1477-7525-9-36. PMID 21600054
- [Derived] Reilly MC, Gooch KL, Wong RL, Kupper H, van der Heijde D. Validity, reliability and responsiveness of the Work Productivity and Activity Impairment Questionnaire in ankylosing spondylitis. Rheumatology (Oxford). 2010 Apr;49(4):812-9. doi: 10.1093/rheumatology/kep457. Epub 2010 Jan 25. PMID 20100797
- [Derived] van der Heijde D, Salonen D, Weissman BN, Landewe R, Maksymowych WP, Kupper H, Ballal S, Gibson E, Wong R; Canadian (M03-606) study group; ATLAS study group. Assessment of radiographic progression in the spines of patients with ankylosing spondylitis treated with adalimumab for up to 2 years. Arthritis Res Ther. 2009;11(4):R127. doi: 10.1186/ar2794. Epub 2009 Aug 24. PMID 19703304
- [Derived] van der Heijde DM, Revicki DA, Gooch KL, Wong RL, Kupper H, Harnam N, Thompson C, Sieper J; ATLAS Study Group. Physical function, disease activity, and health-related quality-of-life outcomes after 3 years of adalimumab treatment in patients with ankylosing spondylitis. Arthritis Res Ther. 2009;11(4):R124. doi: 10.1186/ar2790. Epub 2009 Aug 17. PMID 19686597
- [Derived] van der Heijde D, Schiff MH, Sieper J, Kivitz AJ, Wong RL, Kupper H, Dijkmans BA, Mease PJ, Davis JC Jr; ATLAS Study Group. Adalimumab effectiveness for the treatment of ankylosing spondylitis is maintained for up to 2 years: long-term results from the ATLAS trial. Ann Rheum Dis. 2009 Jun;68(6):922-9. doi: 10.1136/ard.2007.087270. Epub 2008 Aug 13. PMID 18701556
- [Derived] Dougados M, Luo MP, Maksymowych WP, Chmiel JJ, Chen N, Wong RL, Davis JC Jr, van der Heijde D; ATLAS STUDY GROUP. Evaluation of the patient acceptable symptom state as an outcome measure in patients with ankylosing spondylitis: data from a randomized controlled trial. Arthritis Rheum. 2008 Apr 15;59(4):553-60. doi: 10.1002/art.23527. PMID 18383418
- [Derived] van der Heijde D, Pangan AL, Schiff MH, Braun J, Borofsky M, Torre J, Davis JC Jr, Wong RL, Kupper H, Collantes E; ATLAS Study Group. Adalimumab effectively reduces the signs and symptoms of active ankylosing spondylitis in patients with total spinal ankylosis. Ann Rheum Dis. 2008 Sep;67(9):1218-21. doi: 10.1136/ard.2007.082529. Epub 2007 Dec 4. PMID 18056755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with active ankylosing spondylitis (AS) who have an inadequate response or intolerance to 1 or more nonsteroidal antiinflammatory drugs and who may have also failed 1 or more therapies with disease-modifying antirheumatic drugs.
Pre-assignment Details: Subjects were randomized 2:1 to receive either 40 mg adalimumab subcutaneous (sc) every other week (eow) or matched placebo for the 24-week double-blind placebo-controlled period of the study. After 12 weeks, subjects without a reduction of signs and symptoms in ankylosing spondylitis (ASAS 20) were considered for open-label adalimumab treatment.
Groups:
- Adalimumab: Subjects on active treatment received SC injection of 40 mg adalimumab every other week.
- Placebo: Subjects on placebo treatment received SC injection of matched placebo every other week.
- Any Adalimumab: 40 mg every other week (eow), subcutaneous (SC)
Period: Double-Blind Period
Arm/Group | Adalimumab | Placebo | Any Adalimumab
Started | 208 | 107 | 0 (This treatment group is not applicable to the Double-Blind Period.)
Completed | 195 | 101 | 0
Not Completed | 13 | 6 | 0
Not completed — Adverse Event | 5 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Lack/loss of efficacy | 2 | 2 | 0
Not completed — Contemplating pregnancy | 1 | 0 | 0
Not completed — Undiagnosed pre-existing condition | 0 | 1 | 0
Period: Open-Label Period
Arm/Group | Adalimumab | Placebo | Any Adalimumab
Started | 0 (This treatment group is not applicable to the Open-Label Period.) | 0 (This treatment group is not applicable to the Open-Label Period.) | 311 (1 subject who discontinued for personal reasons subsequently died 450 days after last dose.)
Completed | 0 | 0 | 202
Not Completed | 0 | 0 | 109
Not completed — Adverse Event | 0 | 0 | 38
Not completed — Withdrawal by Subject | 0 | 0 | 29
Not completed — Lost to Follow-up | 0 | 0 | 13
Not completed — Lack of Efficacy | 0 | 0 | 15
Not completed — Pregnancy | 0 | 0 | 3
Not completed — Contemplating pregnancy | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Personal reason | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Placebo | Total
Number analyzed (Participants) | 208 | 107 | 315
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 205 | 104 | 309
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.69) | 43.4 (11.32) | 42.2 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 28 | 79
  Male | 157 | 79 | 236
Region of Enrollment [Number; unit: participants]
  United States | 100 | 48 | 148
  Europe | 108 | 59 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders With a Reduction of Signs and Symptoms of Ankylosing Spondylitis (AS) as Measured With ASAS International Working Group Response Criteria (ASAS 20).
Description: ASAS 20 responders - improvement of >=20% and absolute improvement of >=10 units from Baseline in a visual analog scale (VAS) for >=3 of 4 domains; Patient's Global Assessment of disease activity VAS (0 [none]-100 [severe]), Total Back Pain VAS (0 [no pain]-100 [severe]), BASFI VAS (0 [easy]-100[impossible]); and Inflammation VAS (0 [none]-10 [very severe]) and absence of deterioration in the potential remaining domain, defined as a worsening of >=20% and a net worsening of >=10 units. Applied to each scale and not to an overall global scale.
Time Frame: Week 12
Measure: Number; unit: Participants (responders, nonresponders)
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 208 | 107
Participants (responders, nonresponders)
  Responder | 121 | 22
  Nonresponder | 83 | 82
  Missing | 4 | 3
Statistical Analysis 1: Comparison: Adalimumab vs Placebo; ASAS 20 response rates of the adalimumab group were compared with the placebo group using Pearson's Chi-square test. The counts and percentages were calculated for total sample and by therapy group. Statistical tests were 2-sided. For the statistical analysis, subjects with missing data before Week 12 were considered as nonresponders. The comparisons were performed at an alpha level = 0.05; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Difference (RD) = 37.6, 95% CI [27.4 to 47.8] — Risk difference is measured as a percentage

2. Primary Outcome: Mean Change in the Modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) Compared Against a Historical Control Group (Outcomes in Ankylosing Spondylitis International Study [OASIS]) Using the ANCOVA Model Adjusting for Baseline mSASSS Score
Description: Radiographic progression was based on change in mSASSS scoring (comparison of the means) from double-blind Baseline visit to Week 104. The mSASSS is the sum of the lumbar and cervical spine score ( 0 [no change] to 72 [progression]), derived from scoring the anterior site of the lumbar spine (T12 to S1) and the cervical spine (C2 to T1) as either 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), 3 (bridging syndesmophyte), or N (vertebral body not evaluable). Data from NCT00195819 was compared with data from AS patients in OASIS.
Time Frame: Week 104
Population: The OASIS cohort is a historical control group of Dutch, French, and Belgian patients with AS who have been followed up since 1996. These patients participated in a follow-up study on the natural course of AS with conventional (non-biologic) treatment.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Any Adalimumab: By duration of exposure to adalimumab 40 mg every other week, subcutaneous
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 237
score on a scale
  Adalimumab in M03-607 (N = 237) | 0.9 (0.19)
  OASIS (N = 169) | 0.9 (0.23)
Statistical Analysis 1: Comparison: Any Adalimumab; Test type: Superiority or Other; p = 0.985, ANCOVA; Mean Difference (Net) = 0.0, Standard Error of Mean 0.30

3. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Assessments of Ankylosing Spondylitis (ASAS) 20 - Through Week 260 of Adalimumab Exposure
Description: ASAS 20 responders - improvement of >=20% and absolute improvement of >=10 units from Baseline in a visual analog scale (VAS) for >=3 of 4 domains; Patient's Global Assessment of disease activity VAS; (0[none]-100 [severe]), Total Back Pain VAS; (0 [no pain]-100 [severe]), BASFI VAS (0 [easy ]-100[impossible]); and Inflammation VAS (0 [none] to 10 [very severe]) and absence of deterioration in the potential remaining domain, defined as a worsening of >=20% and a net worsening of >=10 units. Applied to each scale and not to an overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: Any Adalimumab Set - includes all participants who received at least 1 dose of adalimumab during the study, in either the double-blind or the open-label phase. 204 participants were randomized to 40 mg adalimumab every other week (eow) and 107 to placebo. The Any Adalimumab Set is analyzed by duration of exposure (weeks) to adalimumab.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 171
  Week 24 Responders (n = 298) | 204
  Week 52 Responders (n = 282) | 198
  Week 76 Responders (n = 269) | 199
  Week 104 Responders (n = 261) | 192
  Week 128 Responders (n = 242) | 181
  Week 156 Responders (n = 234) | 174
  Week 180 Responders (n = 226) | 180
  Week 208 Responders (n = 217) | 172
  Week 220 Responders (n = 210) | 170
  Week 232 Responders (n = 204) | 162
  Week 244 Responders (n = 187) | 153
  Week 260 Responders (n = 125) | 111

4. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Assessments of Ankylosing Spondylitis (ASAS) 50 - Through Week 260 of Adalimumab Exposure
Description: ASAS 50 responders - improvement of >=50% and absolute improvement of >=20 units from Baseline in a visual analog scale (VAS) for >=3 of 4 domains: Patient's Global Assessment of disease activity VAS (0 [none] to 100 [severe]); Total Back Pain VAS (0 [no pain] to 100 [severe]); BASFI VAS (0 [easy] to 100[impossible]); and Inflammation VAS (1 [none] to 10 [very severe]); and absence of deterioration in the potential remaining domain, defined as a worsening of >=20% and a net worsening of >=10 units. Applied to each scale and not to an overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 105
  Week 24 Responders (n = 298) | 122
  Week 52 Responders (n = 282) | 131
  Week 76 Responders (n = 269) | 144
  Week 104 Responders (n = 261) | 144
  Week 128 Responders (n = 242) | 127
  Week 156 Responders (n = 234) | 137
  Week 180 Responders (n = 226) | 131
  Week 208 Responders (n = 217) | 121
  Week 220 Responders (n = 210) | 130
  Week 232 Responders (n = 204) | 125
  Week 244 Responders (n = 187) | 111
  Week 260 Responders (n = 125) | 86

5. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Assessments of Ankylosing Spondylitis (ASAS) 70 - Through Week 260 of Adalimumab Exposure
Description: ASAS 70 responders - improvement of >=70% and absolute improvement of >=30 units from Baseline in a visual analog scale (VAS) for >=3 of 4 domains: Patient's Global Assessment of disease activity VAS (0 [none] to 100 [severe]), Total Back Pain VAS; (0 [no pain] - 100 [severe]), BASFI VAS (0 [easy] to 100[impossible]); and Inflammation VAS (1 [none] to 10 [very severe]); and absence of deterioration in the potential remaining domain, defined as defined as a worsening of >= 20% and a net worsening of >= 10 units. Applied to each scale and not to an overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 62
  Week 24 Responders (n = 298) | 74
  Week 52 Responders (n = 282) | 91
  Week 76 Responders (n = 269) | 99
  Week 104 Responders (n = 261) | 102
  Week 128 Responders (n = 242) | 98
  Week 156 Responders (n = 234) | 97
  Week 180 Responders (n = 226) | 90
  Week 208 Responders (n = 217) | 93
  Week 220 Responders (n = 210) | 87
  Week 232 Responders (n = 204) | 89
  Week 244 Responders (n = 187) | 88
  Week 260 Responders (n = 125) | 69

6. Secondary Outcome: Mean Change in Patient's Global Assessment of Disease Activity in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the effect of adalimumab 40 mg every other week (eow) on patient's global assessment of disease activity. The patient was to assess his/her disease activity in the past week using a visual analog scale (VAS) on a scale of 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mm
  Week 12 (n = 309) | -25.24 (28.029)
  Week 24 (n = 297) | -31.07 (27.663)
  Week 52 (n = 281) | -33.62 (27.803)
  Week 76 (n = 268) | -36.58 (27.425)
  Week 104 (n = 260) | -37.21 (29.090)
  Week 128 (n = 241) | -38.10 (28.778)
  Week 156 (n = 233) | -39.11 (28.510)
  Week 180 (n = 225) | -40.30 (26.378)
  Week 208 (n = 216) | -39.87 (28.222)
  Week 220 (n = 209) | -40.44 (27.913)
  Week 232 (n = 203) | -40.69 (27.205)
  Week 244 (n = 186) | -41.19 (26.962)
  Week 260 (n = 124) | -45.50 (24.849)

7. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Patient's Global Assessment of Disease Activity (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: The patient assesses his/her disease activity for the past week using a Patient Global Assessment of Disease on visual analog scale (VAS) with 0 being none and 100 being severe.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 309) | 192
  Week 24 Responders (n = 297) | 214
  Week 52 Responders (n = 281) | 213
  Week 76 Responders (n = 268) | 211
  Week 104 Responders (n = 260) | 201
  Week 128 Responders (n = 241) | 185
  Week 156 Responders (n = 233) | 184
  Week 180 Responders (n = 225) | 184
  Week 208 Responders (n = 216) | 179
  Week 220 Responders (n = 209) | 175
  Week 232 Responders (n = 203) | 168
  Week 244 Responders (n = 186) | 160
  Week 260 Responders (n = 124) | 112

8. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Functional Index (BASFI) in Subjects With Adalimumab Exposure Through Week 260
Description: BASFI consist of a set of 10 questions designed to determine the degree of functional limitation in subjects with AS. The BASFI score was derived based on the average of questions 1 through 10. The first 8 questions considered activities related to functional anatomy and the final 2 questions assessed the subject's ability to cope with everyday life over the last week. A 100-mm visual analog scale (VAS) was used to answer the questions and the mean of the ten scales gave the BASFI score a value between 0 (easy) and 100 (impossible).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mm
  Week 12 (n = 310) | -16.12 (19.369)
  Week 24 (n = 298) | -20.45 (19.831)
  Week 52 (n = 282) | -22.94 (21.005)
  Week 76 (n = 269) | -25.13 (21.087)
  Week 104 (n = 261) | -26.24 (22.391)
  Week 128 (n = 242) | -26.52 (21.811)
  Week 156 (n = 234) | -27.24 (22.802)
  Week 180 (n = 226) | -28.35 (21.745)
  Week 208 (n = 217) | -27.92 (21.656)
  Week 220 (n = 210) | -27.70 (22.216)
  Week 232 (n = 205) | -28.30 (22.418)
  Week 244 (n = 187) | -29.33 (21.612)
  Week 260 (n = 125) | -31.44 (20.508)

9. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in BASFI (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: BASFI consisted of 10 Visual Analog Scale (VAS) questions with a response ranging from 0 (easy) to 100 (impossible). The BASFI score was derived based on the average of questions 1 through 10. A responder is a subject who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 170
  Week 24 Responders (n = 298) | 190
  Week 52 Responders (n = 282) | 186
  Week 76 Responders (n = 269) | 188
  Week 104 Responders (n = 261) | 189
  Week 128 Responders (n = 242) | 179
  Week 156 Responders (n = 234) | 175
  Week 180 Responders (n = 226) | 177
  Week 208 Responders (n = 217) | 167
  Week 220 Responders (n = 210) | 160
  Week 232 Responders (n = 205) | 159
  Week 244 Responders (n = 187) | 148
  Week 260 Responders (n = 125) | 103

10. Secondary Outcome: Mean Change in Total Back Pain Visual Analog Scale (VAS) in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the effect of 40 mg every other week (eow) adalimumab on Total Back Pain VAS. The subject was to assess his/her disease activity in the past week using a total spine VAS on a scale 0 (no pain) to 100 (severe pain).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mm
  Week 12 (n = 310) | -24.51 (28.334)
  Week 24 (n = 298) | -31.02 (27.323)
  Week 52 (n = 282) | -34.09 (28.646)
  Week 76 (n = 269) | -36.55 (26.897)
  Week 104 (n = 261) | -37.34 (29.839)
  Week 128 (n = 242) | -38.15 (29.172)
  Week 156 (n = 234) | -38.43 (28.667)
  Week 180 (n = 226) | -39.40 (27.830)
  Week 208 (n = 217) | -37.93 (30.306)
  Week 220 (n = 210) | -39.30 (28.996)
  Week 232 (n = 204) | -40.31 (29.449)
  Week 244 (n = 187) | -41.66 (29.196)
  Week 260 (n = 125) | -47.83 (24.636)

11. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Total Back Pain (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: Participants assessed disease activity in the past week using a total spine VAS on a scale 0 (no pain) to 100 (severe pain). A responder is a participant who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 181
  Week 24 Responders (n = 298) | 210
  Week 52 Responders (n = 282) | 208
  Week 76 Responders (n = 269) | 204
  Week 104 Responders (n = 261) | 199
  Week 128 Responders (n = 242) | 188
  Week 156 Responders (n = 234) | 178
  Week 180 Responders (n = 226) | 186
  Week 208 Responders (n = 217) | 172
  Week 220 Responders (n = 210) | 165
  Week 232 Responders (n = 204) | 164
  Week 244 Responders (n = 187) | 157
  Week 260 Responders (n = 125) | 111

12. Secondary Outcome: Mean Change in Inflammation (Mean of BASDAI Questions 5 and 6) in Subjects With Adalimumab Exposure Through Week 260
Description: The inflammation score is the mean of the two morning stiffness-related BASDAI visual analog scale (VAS) scores (items 5 and 6 of the BASDAI): overall level of morning stiffness (0 [none] to 10 [very severe]) and duration of morning stiffness (0 [0 hours] to 10 [2 or more hours]). A decrease in inflammation represents improvement.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
cm
  Week 12 (n = 310) | -2.82 (2.700)
  Week 24 (n = 298) | -3.48 (2.640)
  Week 52 (n = 282) | -3.80 (2.743)
  Week 76 (n = 269) | -3.98 (2.674)
  Week 104 (n = 261) | -4.12 (2.780)
  Week 128 (n = 242) | -4.04 (2.754)
  Week 156 (n = 234) | -3.93 (3.978)
  Week 180 (n = 226) | -4.24 (2.664)
  Week 208 (n = 217) | -4.27 (2.677)
  Week 220 (n = 210) | -4.29 (2.677)
  Week 232 (n = 205) | -4.30 (2.700)
  Week 244 (n = 186) | -4.56 (2.610)
  Week 260 (n = 124) | -4.94 (2.470)

13. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Inflammation (Individual Component of ASAS 20) (Mean of BASDAI Questions 5 and 6) Through Week 260 of Adalimumab Exposure
Description: The inflammation score is the mean of the two morning stiffness-related BASDAI visual analog scale (VAS) scores (items 5 and 6 of the BASDAI): overall level of morning stiffness (0 [none] to 10 [very severe]) and duration of morning stiffness (0 [0 hours] to 10 [2 or more hours]). A decrease in inflammation represents improvement.
  A responder is a participant who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline in inflammation (mean of the BASDAI questions 5 and 6 on scale of 0 [none] to 10 [very severe].
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 198
  Week 24 Responders (n = 298) | 231
  Week 52 Responders (n = 282) | 224
  Week 76 Responders (n = 269) | 221
  Week 104 Responders (n = 261) | 215
  Week 128 Responders (n = 242) | 230
  Week 156 Responders (n = 234) | 192
  Week 180 Responders (n = 226) | 191
  Week 208 Responders (n = 217) | 191
  Week 220 Responders (n = 210) | 182
  Week 232 Responders (n = 205) | 176
  Week 244 Responders (n = 186) | 165
  Week 260 Responders (n = 124) | 114

14. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 20 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 (none) to 10 (very severe). Improvement in BASDAI by 20% was assessed. BASDAI Scoring:
  Measure each item of the BASDAI in centimeters (out of a total of 10) BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 205
  Week 24 Responders (n = 298) | 225
  Week 52 Responders (n = 282) | 218
  Week 76 Responders (n = 269) | 219
  Week 104 Responders (n = 261) | 212
  Week 128 Responders (n = 242) | 202
  Week 156 Responders (n = 234) | 192
  Week 180 Responders (n = 226) | 201
  Week 208 Responders (n = 217) | 190
  Week 220 Responders (n = 210) | 181
  Week 232 Responders (n = 205) | 183
  Week 244 Responders (n = 187) | 170
  Week 260 Responders (n = 124) | 117

15. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. Improvement in BASDAI by 50% was assessed. BASDAI Scoring:
  Measure each item of the BASDAI in centimeters (out of a total of 10) BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 133
  Week 24 Responders (n = 298) | 157
  Week 52 Responders (n = 282) | 169
  Week 76 Responders (n = 269) | 173
  Week 104 Responders (n = 261) | 170
  Week 128 Responders (n = 242) | 155
  Week 156 Responders (n = 234) | 156
  Week 180 Responders (n = 226) | 155
  Week 208 Responders (n = 217) | 147
  Week 220 Responders (n = 210) | 148
  Week 232 Responders (n = 205) | 145
  Week 244 Responders (n = 187) | 135
  Week 260 Responders (n = 124) | 96

16. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 70 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. Improvement in BASDAI by 70% was assessed. BASDAI Scoring:
  Measure each item of the BASDAI in centimeters (out of a total of 10) BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 80
  Week 24 Responders (n = 298) | 103
  Week 52 Responders (n = 282) | 113
  Week 76 Responders (n = 269) | 114
  Week 104 Responders (n = 261) | 129
  Week 128 Responders (n = 242) | 115
  Week 156 Responders (n = 234) | 119
  Week 180 Responders (n = 226) | 110
  Week 208 Responders (n = 217) | 113
  Week 220 Responders (n = 210) | 109
  Week 232 Responders (n = 205) | 110
  Week 244 Responders (n = 187) | 104
  Week 260 Responders (n = 124) | 76

17. Secondary Outcome: Mean Change in BASDAI in Subjects With Adalimumab Exposure Through Week 260
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 (none) to 10 (severe). A decrease in BASDAI represents improvement. BASDAI Scoring: 1) Measure each item of the BASDAI in centimeters (out of a total of 10) 2) BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
cm
  Week 12 (n = 310) | -2.38 (2.377)
  Week 24 (n = 298) | -2.90 (2.418)
  Week 52 (n = 282) | -3.16 (2.547)
  Week 76 (n = 269) | -3.38 (2.384)
  Week 104 (n = 261) | -3.54 (2.519)
  Week 128 (n = 242) | -3.53 (2.421)
  Week 156 (n = 234) | -3.45 (3.491)
  Week 180 (n = 226) | -3.79 (2.349)
  Week 208 (n = 217) | -3.78 (2.352)
  Week 220 (n = 210) | -3.73 (2.350)
  Week 232 (n = 205) | -3.79 (2.395)
  Week 244 (n = 187) | -4.08 (2.248)
  Week 260 (n = 124) | -4.44 (2.227)

18. Secondary Outcome: Mean Change in C-Reactive Protein (CRP) (mg/dL) in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the mean changes in CRP in subjects with adalimumab exposure from Baseline through 5 years. The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation via the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation. A decrease in CRP indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mg/dL
  Week 12 (n = 308) | -1.27 (2.092)
  Week 24 (n = 294) | -1.24 (2.275)
  Week 52 (n = 279) | -1.30 (2.221)
  Week 76 (n = 264) | -1.35 (2.314)
  Week 104 (n = 258) | -1.45 (2.333)
  Week 128 (n = 238) | -1.36 (2.589)
  Week 156 (n = 230) | -1.46 (2.604)
  Week 180 (n = 224) | -1.54 (2.530)
  Week 208 (n = 215) | -1.54 (2.740)
  Week 220 (n = 207) | -1.50 (2.956)
  Week 232 (n = 203) | -1.57 (2.709)
  Week 244 (n = 186) | -1.58 (2.748)
  Week 260 (n = 123) | -1.67 (2.623)

19. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured in Assessments of Ankylosing Spondylitis (ASAS) 40 - Through Week 260 of Adalimumab Exposure
Description: ASAS 40 responders - improvement of >=40% and absolute improvement of >=20 units from Baseline in a visual analog scale (VAS) for >=3 of 4 domains; Patient's Global Assessment of disease activity VAS (0 [none] to 100 [severe]); Total Back Pain VAS (0 [no pain] to 100 [severe]); BASFI VAS (0 [easy] to 100[impossible]); and Inflammation VAS (1 [none] to 10 [very severe]); and absence of any deterioration in the potential remaining domain. Applied to each scale and not to an overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 115
  Week 24 Responders (n = 298) | 144
  Week 52 Responders (n = 282) | 143
  Week 76 Responders (n = 269) | 157
  Week 104 Responders (n = 261) | 155
  Week 128 Responders (n = 242) | 140
  Week 156 Responders (n = 234) | 147
  Week 180 Responders (n = 226) | 143
  Week 208 Responders (n = 217) | 131
  Week 220 Responders (n = 210) | 134
  Week 232 Responders (n = 204) | 134
  Week 244 Responders (n = 187) | 118
  Week 260 Responders (n = 125) | 88

20. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured in Assessments of Ankylosing Spondylitis Ankylosing Spondylitis (ASAS) 5/6 in Subjects With Adalimumab Exposure Through Week 260
Description: The change in ASAS 5/6 was evaluated for the effect of adalimumab on structural damage.
  ASAS 5/6 criteria is the 20% improvement in 5 out of 6 domains (physical function [BASFI], Total Back Pain, Patient's Global Assessment of Disease Activity, Inflammation [mean of Questions 5 and 6 of the BASDAI], spinal mobility [BASMI], and acute phase reactants [CRP]).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 309) | 145
  Week 24 Responders (n = 297) | 184
  Week 52 Responders (n = 281) | 169
  Week 76 Responders (n = 268) | 179
  Week 104 Responders (n = 260) | 177
  Week 128 Responders (n = 241) | 159
  Week 156 Responders (n = 232) | 157
  Week 180 Responders (n = 225) | 160
  Week 208 Responders (n = 216) | 152
  Week 220 Responders (n = 208) | 148
  Week 232 Responders (n = 203) | 144
  Week 244 Responders (n = 186) | 132
  Week 260 Responders (n = 125) | 95

21. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured by ASAS Partial Remission Response in Subjects With Adalimumab Exposure Through Week 260
Description: ASAS partial remission was calculated as follows: A value below 20 on a 0 - 100 point scale in each of the four domains of the ASAS (Patient's Global Assessment of Disease Activity, Pain, Function, and Inflammation). Partial remission is also regarded as a low disease activity state.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 Responders (n = 310) | 62
  Week 24 Responders (n = 298) | 75
  Week 52 Responders (n = 282) | 94
  Week 76 Responders (n = 269) | 101
  Week 104 Responders (n = 261) | 100
  Week 128 Responders (n = 242) | 97
  Week 156 Responders (n = 234) | 96
  Week 180 Responders (n = 226) | 87
  Week 208 Responders (n = 217) | 86
  Week 220 Responders (n = 210) | 78
  Week 232 Responders (n = 204) | 96
  Week 244 Responders (n = 186) | 74
  Week 260 Responders (n = 124) | 63

22. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Metrology Index (BASMI) in Subjects With Adalimumab Exposure Through Week 260
Description: BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. BASMI 0 = indicates mild disease involvement, 1 = moderate disease, and 2 = severe disease involvement. The results for cervical rotation and lumbar side flexion are the means of the left and right measurements. Scoring range 0-10. The higher the BASMI score, the more severe was the subject's limitation of movement due to their AS.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 309) | -0.43 (1.313)
  Week 24 (n = 294) | -0.60 (1.397)
  Week 52 (n = 282) | -0.73 (1.375)
  Week 76 (n = 268) | -0.77 (1.400)
  Week 104 (n = 261) | -0.70 (1.502)
  Week 128 (n = 242) | -0.67 (1.442)
  Week 156 (n = 233) | -0.80 (1.472)
  Week 180 (n = 225) | -0.70 (1.530)
  Week 208 (n = 215) | -0.75 (1.535)
  Week 220 (n = 208) | -0.74 (1.592)
  Week 232 (n = 201) | -0.71 (1.579)
  Week 244 (n = 187) | -0.68 (1.500)
  Week 260 (n = 124) | -0.76 (1.521)

23. Secondary Outcome: Mean Change in Chest Expansion (CE) in Subjects With Adalimumab Exposure Through Week 260 [
Description: The patient is in a sitting position on the examination table with the hands on the hips. A pen mark is made at the xiphisternum and a tape measure placed around the circumference of the patient's chest at this level. The patient is asked to take a deep breath and to exhale as completely as possible while looking directly ahead. The measurement (in cm) is noted. The patient is asked to inhale as deeply as possible and the measurement (in cm) is noted. The difference in the 2 measurement points (in cm) constitutes the value for CE.
  An increase in chest expansion represents improvement
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
cm
  Week 12 (n = 277) | 0.34 (1.570)
  Week 24 (n = 237) | 0.25 (1.445)
  Week 52 (n = 234) | 0.71 (6.574)
  Week 104 (n = 261) | 0.59 (1.632)
  Week 128 (n = 199) | 1.24 (7.627)
  Week 156 (n = 230) | 0.58 (1.722)
  Week 180 (n = 184) | 0.42 (1.865)
  Week 208 (n = 202) | 0.96 (5.877)
  Week 220 (n = 61) | 0.86 (1.962)
  Week 232 (n = 142) | 0.60 (2.657)
  Week 244 (n = 61) | 2.61 (15.450)
  Week 260 (n = 123) | 1.25 (9.479)

24. Secondary Outcome: Mean Change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) in Subjects With Adalimumab Exposure Through Week 260
Description: MASES is measured by scoring of entheses of 0 (no tenderness) to 3 (severe tenderness) at 13 sites on the body. The score was derived as the sum of the 13 scores divided by 3 and the total range is 0 to 13 (minimum to maximum number and severity of enthesitis).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 308) | -2.25 (5.888)
  Week 24 (n = 294) | -2.97 (5.924)
  Week 52 (n = 279) | -3.28 (5.908)
  Week 76 (n = 226) | -3.27 (5.864)
  Week 104 (n = 259) | -3.43 (6.560)
  Week 128 (n = 201) | -3.18 (6.043)
  Week 156 (n = 229) | -3.28 (6.154)
  Week 180 (n = 184) | -3.44 (5.699)
  Week 208 (n = 214) | -3.38 (6.070)
  Week 232 (n = 170) | -3.25 (5.718)
  Week 260 (n = 167) | -4.06 (6.528)

25. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Global Index (BAS-G) in Subjects With Adalimumab Exposure Through Week 260
Description: BAS-G was measured by two VAS scores (0 to 100 mm) to reflect the effect of Ankylosing Spondylitis on subject's well-being over the past week and over the last 6 months, respectively. The average of these two scores was reported.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 Responders (n = 309) | -20.55 (22.143)
  Week 24 Responders (n = 293) | -29.74 (24.558)
  Week 52 Responders (n = 281) | -35.48 (25.949)
  Week 76 Responders (n = 269) | -39.29 (25.817)
  Week 104 Responders (n = 261) | -40.36 (27.532)
  Week 128 Responders (n = 242) | -41.47 (26.244)
  Week 156 Responders (n = 234) | -40.66 (26.834)
  Week 180 Responders (n = 226) | -42.59 (25.816)
  Week 208 Responders (n = 217) | -42.21 (26.698)
  Week 220 Responders (n = 209) | -41.85 (26.493)
  Week 232 Responders (n = 205) | -41.59 (26.898)
  Week 244 Responders (n = 187) | -44.86 (25.016)
  Week 260 Responders (n = 125) | -47.66 (24.845)

26. Secondary Outcome: Mean Change in Swollen Joint Count for 44 Joints (44 SJC) in Subjects With Adalimumab Exposure Through Week 260
Description: Change from Baseline in the swollen joint index. An assessment of 44 joints for SJC done by physical examination. Joint swelling was classified as present ("1"), absent ("0") or injected/replaced ("9"). The joints assessed were: Sternoclavicular, Acromioclavicular, Shoulder, Elbow, Wrist, Metacarpophalangeal (1-5), Thumb interphalangeal, Proximal interphalangeal (2-5, Knee, Ankle, and Metatarsophalangeal (1-5).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 311) | -0.18 (3.280)
  Week 24 (n = 295) | -0.40 (2.608)
  Week 52 (n = 281) | -0.36 (3.360)
  Week 76 (n = 231) | -0.59 (3.044)
  Week 104 (n = 261) | -0.60 (3.723)
  Week 128 (n = 200) | -0.79 (3.434)
  Week 156 (n = 231) | -0.60 (3.446)
  Week 180 (n = 187) | -0.69 (3.669)
  Week 208 (n = 215) | -0.54 (4.412)
  Week 232 (n = 170) | -0.74 (3.822)
  Week 260 (n = 169) | -0.70 (3.863)

27. Secondary Outcome: Mean Change From Baseline in the Tender Joint Count for 46 Joints (TJC 46) in Subjects With Adalimumab Exposure Through Week 260
Description: Assessment of 46 joints for TJC was done by physical examination. Joint tenderness was classified as present ("1"), absent ("0") or injected/replaced ("9"). The joints assessed were: Sternoclavicular, Acromioclavicular, Shoulder, Elbow, Wrist, Metacarpophalangeal (1-5), Thumb interphalangeal, Proximal interphalangeal (2-5, Hip, Knee, Ankle, and Metatarsophalangeal (1-5).
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 311) | -1.09 (5.193)
  Week 24 (n = 295) | -1.41 (5.297)
  Week 52 (n = 281) | -1.70 (6.330)
  Week 76 (n = 231) | -1.87 (6.007)
  Week 104 (n = 261) | -2.22 (6.816)
  Week 128 (n = 202) | -2.16 (6.161)
  Week 156 (n = 233) | -2.28 (5.361)
  Week 180 (n = 187) | -2.88 (5.358)
  Week 208 (n = 215) | -2.44 (5.270)
  Week 232 (n = 171) | -2.76 (5.402)
  Week 260 (n = 169) | -2.63 (6.348)

28. Secondary Outcome: Mean Change in Physician's Global Assessment of Disease Activity in Subjects With Adalimumab Exposure Through Week 260
Description: The physician will globally assess the subject's current disease state using a 100-mm VAS scale with 0 being very good and 100 being very bad.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mm
  Week 12 Responders (n = 310) | -24.36 (26.877)
  Week 24 Responders (n = 297) | -29.69 (27.662)
  Week 52 Responders (n = 281) | -34.01 (26.066)
  Week 76 Responders (n = 267) | -37.16 (23.291)
  Week 104 Responders (n = 260) | -37.58 (25.726)
  Week 128 Responders (n = 239) | -38.17 (26.787)
  Week 156 Responders (n = 233) | -38.10 (25.726)
  Week 180 Responders (n = 225) | -39.76 (23.903)
  Week 208 Responders (n = 215) | -39.30 (24.764)
  Week 220 Responders (n = 209) | -39.44 (24.361)
  Week 232 Responders (n = 203) | -38.46 (25.529)
  Week 244 Responders (n = 186) | -43.14 (22.824)
  Week 260 Responders (n = 124) | -43.83 (19.383)

29. Secondary Outcome: Mean Change in Nocturnal Pain in Subjects With Adalimumab Exposure Through Week 260
Description: The subject was to assess his/her nocturnal pain intensity for the past week using a Nocturnal Pain Visual Analog Scale (Nocturnal Pain VAS). The range was 0 to 100 mm with no pain being indicated by 0 and worse possible pain by 100.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
mm
  Week 12 (n = 309) | -24.29 (29.281)
  Week 24 (n = 297) | -30.85 (28.473)
  Week 52 (n = 281) | -33.91 (30.280)
  Week 76 (n = 268) | -37.17 (27.931)
  Week 104 (n = 260) | -36.71 (30.261)
  Week 128 (n = 241) | -37.52 (30.796)
  Week 156 (n = 233) | -37.33 (29.194)
  Week 180 (n = 225) | -38.68 (29.810)
  Week 208 (n = 216) | -37.62 (30.925)
  Week 220 (n = 209) | -38.43 (30.946)
  Week 232 (n = 203) | -39.53 (30.433)
  Week 244 (n = 186) | -40.73 (30.098)
  Week 260 (n = 124) | -45.19 (26.944)

30. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Physical Component Summary (PCS) Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0 (no functioning) to 100 (highest level of functioning). The SF-36 Health Survey Index was completed by participants. Components of the SF-36 included the PCS and MCS, respectively. An increase in SF-36 PCS or MCS indicated improvement.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 278) | 6.92 (8.764)
  Week 24 (n = 237) | 7.30 (8.678)
  Week 52 (n = 278) | 9.07 (9.629)
  Week 76 (n = 227) | 9.70 (9.812)
  Week 104 (n = 256) | 9.95 (10.646)
  Week 128 (n = 196) | 10.01 (10.394)
  Week 156 (n = 230) | 11.23 (9.998)
  Week 180 (n = 184) | 10.67 (9.918)
  Week 208 (n = 214) | 10.39 (10.214)
  Week 232 (n = 168) | 10.76 (9.892)
  Week 260 (n = 165) | 11.83 (9.907)

31. Secondary Outcome: Number of Subjects With SF-36 Physical Component Summary (PCS) of Minimal Clinically Important Difference (MCID) Response Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0(no functioning) to 100 (highest level of functioning).
  Responders were subjects whose change in PCS score fulfilled the Minimal Clinically Important Difference (MCID). The MCID for PCS was determined by a >= 3.0 point increase during exposure to adalimumab.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 (n = 278) | 178
  Week 24 (n = 237) | 162
  Week 52 (n = 278) | 198
  Week 76 (n = 227) | 166
  Week 104 (n = 256) | 194
  Week 128 (n = 196) | 141
  Week 156 (n = 230) | 186
  Week 180 (n = 184) | 138
  Week 208 (n = 214) | 156
  Week 232 (n = 168) | 130
  Week 260 (n = 165) | 129

32. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Mental Component Summary (MCS) Through Week 260 of Adalimumab Exposure
Description: as for outcome 30
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 278) | 3.18 (11.114)
  Week 24 (n = 237) | 4.24 (9.757)
  Week 52 (n = 278) | 4.56 (10.404)
  Week 76 (n = 227) | 4.31 (10.907)
  Week 104 (n = 256) | 4.42 (11.466)
  Week 128 (n = 196) | 3.71 (10.519)
  Week 156 (n = 230) | 4.19 (11.551)
  Week 180 (n = 184) | 4.64 (11.056)
  Week 208 (n = 214) | 5.50 (10.760)
  Week 232 (n = 168) | 4.66 (10.131)
  Week 260 (n = 165) | 5.74 (10.758)

33. Secondary Outcome: Number of Subjects With SF-36 Mental Component Summary (MCS) of Minimal Clinically Important Difference (MCID) Response Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0(no functioning) to 100 (highest level of functioning).
  Responders were subjects whose change in MCS fulfilled the Minimal Clinically Important Difference (MCID). The MCID for MCS was determined by a >= 3.0 point increase during exposure to adalimumab.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 (n = 278) | 132
  Week 24 (n = 237) | 121
  Week 52 (n = 278) | 137
  Week 76 (n = 227) | 120
  Week 104 (n = 256) | 132
  Week 128 (n = 196) | 100
  Week 156 (n = 230) | 115
  Week 180 (n = 184) | 94
  Week 208 (n = 214) | 116
  Week 232 (n = 168) | 88
  Week 260 (n = 165) | 97

34. Secondary Outcome: Mean Change in Health Utilities Index-3 (HUI-3) Through Week 260 of Adalimumab Exposure
Description: The HUI-3 is a generic approach to the measurement of health status and assessment of health-related quality of life (HRQL). The HUI-3 classification is comprised of a total score and 8 attributes - Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition and Pain. The attributes are measures on a scale from the worst score of 0 to best score of 1. The total score scale ranges from dead (= 0) and perfect health (= 1). The total score can have a negative score that is interpreted as worse than dead and the lower limit is -0.36. An increase in the HUI-3 score represents improvement.
Time Frame: Baseline, Weeks 24, 52, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 24 (n = 303) | 0.18 (0.245)
  Week 52 (n = 239) | 0.20 (0.258)
  Week 104 (n = 263) | 0.20 (0.258)
  Week 128 (n = 201) | 0.20 (0.245)
  Week 156 (n = 232) | 0.22 (0.274)
  Week 180 (n = 187) | 0.22 (0.245)
  Week 208 (n = 216) | 0.22 (0.244)
  Week 232 (n = 171) | 0.23 (0.247)
  Week 260 (n = 166) | 0.26 (0.244)

35. Secondary Outcome: Mean Change in the Ankylosing Spondylitis Quality of Life Questionaire (ASQoL) in Subjects Through Week 260 of Adalimumab Exposure
Description: ASQoL determined participants' quality of life and is comprised of 18 questions (yes or no) to be completed by the participant. Each statement on the ASQoL is given a score of "1" or "0." All item scores were summed to give a total score or index. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement.
Time Frame: Baseline, Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
score on a scale
  Week 12 (n = 284) | -3.26 (4.144)
  Week 24 (n = 242) | -3.69 (4.081)
  Week 52 (n = 281) | -4.29 (4.475)
  Week 76 (n = 232) | -4.36 (4.383)
  Week 104 (n = 261) | -4.80 (4.497)
  Week 128 (n = 202) | -4.59 (4.501)
  Week 156 (n = 233) | -5.05 (4.630)
  Week 180 (n = 186) | -4.95 (4.526)
  Week 208 (n = 217) | -5.18 (4.406)
  Week 232 (n = 173) | -5.09 (4.052)
  Week 260 (n = 169) | -5.66 (4.188)

36. Secondary Outcome: Number of Subjects With Ankylosing Spondylitis Quality of Life Questionaire (ASQoL) MCID Response (MCID <= -1.8 Points) Through Week 260 of Adalimumab Exposure
Description: ASQoL determined participants' quality of life and is comprised of 18 questions (yes or no) to be completed by the participant. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement. Responders are participants with a minimal clinically important difference (MCID) <= -1.8 points. MCID was determined by a >= 1.8 score decrease during exposure to adalimumab.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 (n = 284) | 176
  Week 24 (n = 242) | 160
  Week 52 (n = 281) | 204
  Week 76 (n = 232) | 170
  Week 104 (n = 261) | 198
  Week 128 (n = 202) | 151
  Week 156 (n = 233) | 179
  Week 180 (n = 186) | 144
  Week 208 (n = 217) | 169
  Week 232 (n = 173) | 139
  Week 260 (n = 169) | 142

37. Secondary Outcome: Number of Subjects Achieving the Patient Acceptable Symptoms State Through Week 260 of Adalimumab Exposure
Description: Completed by subject at each visit. The Patient Acceptable Symptoms State (PASS) was a participant-reported outcome where participants were expected to respond (yes/no) to the following question:
  Considering all the different ways your disease is affecting you, if you would stay in this state for the next months, do you consider that your current state is satisfactory?
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 311
participants
  Week 12 (n = 310) | 140
  Week 24 (n = 298) | 153
  Week 52 (n = 282) | 164
  Week 76 (n = 269) | 162
  Week 104 (n = 259) | 172
  Week 128 (n = 194) | 124
  Week 156 (n = 230) | 161
  Week 180 (n = 185) | 127
  Week 208 (n = 212) | 144
  Week 232 (n = 172) | 122
  Week 260 (n = 165) | 112

ADVERSE EVENTS:
Time Frame: Baseline through 260 weeks of adalimumab exposure
Groups:
- Any Adalimumab: By duration of exposure to any adalimumab 40 mg eow, subcutaneous
Arm/Group | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 96/311
Other Adverse Events (participants affected / at risk) | 279/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Adalimumab (N=311)
Aortic valve incompetence (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 1
Inner ear disorder (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Enterocele (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Oesophageal hypomotility (Gastrointestinal disorders) | 1
Oesophageal rupture (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 5
Injection site reaction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 2
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Cellullitis (Infections and infestations) | 3
Endocarditis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Device failure (Injury, poisoning and procedural complications) | 1
Electric shock (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Nerve injury (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 2
Stent occlusion (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periathritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Breast enlargement (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Abortion induced (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Adalimumab (N=311)
Iritis (Eye disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 41
Nausea (Gastrointestinal disorders) | 30
Fatigue (General disorders) | 37
Injection site reaction (General disorders) | 16
Oedema peripheral (General disorders) | 19
Pain (General disorders) | 18
Pyrexia (General disorders) | 27
Seasonal allergy (Immune system disorders) | 19
Bronchitis (Infections and infestations) | 41
Gastroenteritis (Infections and infestations) | 17
Influenza (Infections and infestations) | 38
Nasopharyngitis (Infections and infestations) | 110
Pharyngitis (Infections and infestations) | 23
Rhinitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 47
Upper respiratory tract infection (Infections and infestations) | 77
Viral infection (Infections and infestations) | 28
Contusion (Injury, poisoning and procedural complications) | 18
Alanine aminotransferase increased (Investigations) | 20
Hypercholesterolaemia (Metabolism and nutrition disorders) | 25
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 54
Back pain (Musculoskeletal and connective tissue disorders) | 38
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24
Tendonitis (Musculoskeletal and connective tissue disorders) | 17
Dizziness (Nervous system disorders) | 22
Headache (Nervous system disorders) | 60
Paraesthesia (Nervous system disorders) | 17
Anxiety (Psychiatric disorders) | 20
Depression (Psychiatric disorders) | 22
Insomnia (Psychiatric disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 44
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 18
Eczema (Skin and subcutaneous tissue disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 19
Psoriasis (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 27
Hypertension (Vascular disorders) | 45

LIMITATIONS AND CAVEATS:
Interim results are shown for subjects after 12 weeks for efficacy parameters and 24 weeks for safety parameters. Subjects who discontinued the study before Week 12 and subjects with missing values were classified as nonresponders for efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.